CLINICAL TRIAL: NCT02346669
Title: Fecal Microbiota Transplantation for Diabetes Mellitus Type II in Obese Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TASMC-14-NM-447-CTIL
Record Dates: First submitted 2015-01-08; First posted 2015-01-27 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
Keywords: Microbiota; Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Gastroscopy; Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- FMT from a lean donor+ high fat diet (Active Comparator): Patients will undergo FMT (Fecal Microboita Transplantation) from a lean donor twice during study through a gastroscopy:
  1. at time 0
  2. after 6 weeks Patient will start high fat low fiber diet 2 weeks before first FMT and continue on consuming the same diet 9 weeks after the first FMT. Patient will be followed up by a nutritionist through the the study.
  Interventions: Procedure: gastroscopy; Drug: Fecal Microbiota Transplantation; Other: high fat low fiber diet
- FMT from a lean donor+ sham diet (Sham Comparator): Patients will undergo FMT (Fecal Microboita Transplantation) from a lean donor twice during study through a gastroscopy:
  1. at time 0
  2. after 6 weeks Patient will start sham diet (no change in fat/fiber consumption) 2 weeks before first FMT and continue on consuming the same diet 9 weeks after the first FMT. Patient will be followed up by a nutritionist through the the study.
  Interventions: Procedure: gastroscopy; Drug: Fecal Microbiota Transplantation; Other: sham diet
- FMT from lean donor+ low fat diet (Active Comparator): Patients will undergo FMT (Fecal Microboita Transplantation) from a lean donor twice during study through a gastroscopy:
  1. at time 0
  2. after 6 weeks Patient will start low fat high fiber diet 2 weeks before first FMT and continue on consuming the same diet 9 weeks after the first FMT. Patient will be followed up by a nutritionist through the the study.
  Interventions: Procedure: gastroscopy; Drug: Fecal Microbiota Transplantation; Other: low fat high fiber diet

INTERVENTIONS:
Procedure: gastroscopy — as detailed in arm description
Drug: Fecal Microbiota Transplantation — as detailed in arm description
Other: high fat low fiber diet — as detailed in arm description
  Arms: FMT from a lean donor+ high fat diet
Other: sham diet — as detailed in arm description
  Arms: FMT from a lean donor+ sham diet
Other: low fat high fiber diet — as detailed in arm description
  Arms: FMT from lean donor+ low fat diet

SUMMARY:
The incidence of obesity has dramatically increased during the last three decades, leading to a significant increase of obesity-related morbidity, including type 2 diabetes mellitus (T2DM) that is characterized by resistance of target tissues to insulin action. T2DM obese patients may be treated by medications or by bariatric surgery. Both alternatives have limitations due to incomplete resolution of the diseases, high cost or potential procedural related morbidity. An increasing body of evidence points to a role of the enteric microbiota in the pathogenesis of obesity-related insulin resistance. In addition to that, the gut microbiota is directly affected by the diet composition. Studies in T2DM mice carrying human gut germs, demonstrated special interactions between the gut microbiota and the host, creating a typical microbiota composition which changes significantly following diet change from a western diet, rich with sugar, to a vegetarian diet rich with fibers. This rapid alternations in the microbiota composition has also shown in humans, after changing from western to high fiber diet. A change in diet life style may lead to an improvement in T2DM symptoms such as decrease in visceral adipose tissue.

DETAILED DESCRIPTION:
Study design:

30 Patients will undergo 2 FMT's from a lean donor and will be randomized into 3 types of diet groups:

1. low fat high fiber diet (20% fat)
2. no change in fat intake (sham diet)
3. high fat low fiber diet (40-45% fat)

The treating physicians and the patients will be blinded for the diet arm. Before and after FMT, patients will be assessed after an overnight fast (and before taking medications) for weight, anthropometric measures, questionnaires (dietary, general health, antibiotic and probiotic exposure, oral diabetes medication quantity, and other drug exposure), blood and stool.

The investigators hypothesize that fecal microbial transplantation from a lean donor to T2DM obese patients, with the combination of low fat high fiber diet, will alter the gut microbiota composition to decrease insulin resistance through microbiota dependent metabolic and immunologic effects.

ELIGIBILITY:
Inclusion Criteria:

* 30≤BMI
* A diagnosis of T2DM (≥3 months) and one of the following:

  1. Fasting glucose level≥126mg/dL and/ or
  2. A stable dose of anti-diabetic drugs for ≥2 weeks and/or
  3. HbA1C≥6.5
* Access to a smart phone supporting the research application for tracking food consumption.

Exclusion Criteria:

* participation in other clinical trial
* incapable of signing an informed consent
* pregnancy or breast feeding
* Antibiotic treatment within the prior 3 months or predicted antibiotic treatment
* insulin medications
* drugs or alcohol addiction
* immune mediated diseases
* type 1 diabetes and latent autoimmune diabetes of adults
* systemic disease
* ischemic heart disease
* probiotics consumption
* a new or unstable treatment with anti diabetic medications

Patients will also be excluded if:

* treated by systemic antibiotic during the study
* will not be compliant with the diet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
30% decrease in insulin resistance | 6 weeks after first FMT
  Lean donor FMT will result in 30% decrease in insulin resistance that will be further enhanced after a second FMT. These will be meditated by an alteration of intestinal microbiota
40% decrease in insulin resistance compared to baseline | 12 weeks after second FMT

SECONDARY OUTCOMES:
Decreased use of diabetes medications | Week 6 and 12 post FMT
Improvement in anthropometric measures and in metabolic indices | week 6 and 12 post FMT
  At least 5% decrease in waist to hip ratio and in total body weight
Maintenance of an improved insulin resistance | 28 weeks post FMT
  Insulin resistance at 28 weeks will be in the range (+5% to -5%) of the value achieved at week 12.
Maintenance of altered of enteric microbiota in the three diet groups | 6, 12, 28 weeks post FMT

CONTACTS AND LOCATIONS:
Overall Officials: Nitsan Maharshak, MD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Department of Gastroentherology, Tel Aviv, Israel